Statistical Analysis Plan I5F-IE-JSCA (v2.0)

Phase 1 Study of IMC-CS4, a Monoclonal Antibody Targeted to the CSF-1 Receptor (CSF-1R), In Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy is Available

NCT01346358

Approval Date: 19-Oct-2012

# 1 Title Page

# Statistical Analysis Plan for Clinical Study

# CP24-1001

Phase 1 Study of IMC-CS4, a Monoclonal Antibody Targeted to the CSF-1 Receptor (CSF-1R), in Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy is Available

IMC-CS4 (LY3022855)

**Indication: Solid tumor** 

This open-label, dose-escalation, Phase 1 study will investigate up to 5 dose levels and enroll approximately 24 subjects (if no dose-limiting toxicity [DLT] is observed). The study will evaluate weekly IMC-CS4 in subjects with advanced solid tumors that are refractory to standard therapy or for which no standard therapy is available and assess the MTD.

ImClone LLC, a wholly-owned subsidiary of Eli Lilly and company (ImClone)
Protocol CP24-1001 (I5F-IE-JSCA)
Phase 1
SAP Version 2.0

## **Confidential Information**

The information contained in this Statistical Analysis Plan (SAP) is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

Approval Date: 19-Oct-2012 GMT

# **2** Table of Contents

| Section | Page |
|-----------------------------------------------------|------|
| 1 Title Page | 1 |
| 2 Table of Contents | |
| 3 Revision history | 3 |
| 3.1 Introduction | 3 |
| 3.2 Revision history | 3 |
| 4 Study Objectives | 4 |
| 4.1 Primary Objective | |
| 4.2 Secondary Objectives | |
| 4.3 Exploratory Objectives | |
| 5 A Priori Statistical Methods | |
| 5.1 Study populations | |
| 5.1.1 All Enrolled Patients | |
| 5.1.2 Safety Population | |
| 5.1.3 Maximum Tolerated Dose (MTD) Population | |
| 5.2 Definitions and data handling conventions | |
| 5.2.1 Safety Data Handling and Definitions | |
| Table 1: Planned Weekly Dose | |
| Table 2: General Dose Reduction Guidelines | |
| 5.2.2 Efficacy Data Handling and Definitions | |
| 5.2.3 General Data Handling | |
| 5.3 Data analysis 5.3.1 Disposition of Patients | |
| 5.3.2 Demographic and Baseline Characteristics | |
| 5.3.3 Analysis of Efficacy Data | 12 |
| 5.3.4 Analysis of Efficacy Data | |
| 5.3.5 Other Assessments or Analyses | |
| 5.4 Interim analyses and data monitoring committees | |
| 5.5 Changes in planned analyses from the protocol | |
| 6 Planned summary tables and Listings | |
| 6.1 Planned Demographic Tables | |
| 6.2 Planned Efficacy Tables | |
| 6.3 Planned Safety Tables | |
| 6.4 Planned Patient Data Listings | |
| Appendix 1: List of Abbreviations | |
| Annandiy 7: Pafarancas | 25 |

# 3 Revision history

#### 3.1 Introduction

This statistical analysis plan for protocol CP24-1001 (I5F-IE-JSCA), Version 3.0, dated 28 March 2012, describes the detailed procedures for executing the planned statistical analyses for the clinical study report. Pharmacokinetic, pharmacodynamic and immunogenicity data will be analyzed by the ImClone LLC Clinical Pharmacology department.

The statistical analyses will be conducted by ImClone LLC or a contract research organization (CRO) using SAS® software Version 9.1.3 or higher.

## 3.2 Revision history

The SAP Version 1.0 was approved prior to First Patient Visit (FPV).

## 4 Study Objectives

## 4.1 Primary Objectives

The primary objectives of this study are to establish the safety profile and characterize the pharmacokinetic profile of IMC-CS4 in the treatment of subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy is available. to determine the maximum tolerated dose (MTD) of IMC-CS4 in the treatment of subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy is available.

## 4.2 Secondary Objectives

The secondary objectives of this study are:

- To define the recommended Phase 2 dose (RP2D);
- To describe the pharmacokinetics (PK) of IMC-CS4; To characterize the pharmacodynamic profile of INC-CS4;
- To assess the pharmacodynamic impact of IMC-CS4 on circulating CSF-1;
- To assess the development of antibodies against IMC-CS4 (immunogenicity); and
- To assess the antitumor activity of IMC-CS4 as monotherapy in the treatment of advanced solid tumors.

#### 4.3 Exploratory Objectives

The exploratory objectives of this study are:

- To assess the pharmacodynamic impact of IMC-CS4 on selected RNA, protein, and circulating markers; and response markers including, but not limited to, CFS-1, soluble CSF-1R and interleukin-34 (IL-34)
- To investigate potential correlation between selected biomarkers and the safety and efficacy of IMC-CS4. To assess the impact of IMC-CS4 monotherapy on LDH, CK, and alkaline phosphatase (AP) isoenymes;

IMC-CS4 (LY3022855)

- To assess the pharmacodynamic impact of IMC-CS-4 on selected cellular and molecular markers to establish a potential correlation with safety and anti-tumor activity
- To assess the pharmacodynamic impact of IMC-CS-4 on various components of the monocyte-macrophage system in hematologic or tissue specimens
- To assess the impacot of IMC-CS4 monotherapy on bone metabolism; and
- To assess the antitumor activity of IMC-CS4 as monotherapy in the treatment of advanced solid tumors.

#### 5 A Priori Statistical Methods

#### 5.1 Study populations

Subjects meeting the inclusion criteria and the exclusion criteria as specified in the study protocol are eligible for enrollment in this study.

#### **5.1.1** All Enrolled Patients

Anyone who signed the informed consent will be included in this population.

## **5.1.2 Safety Population**

All enrolled subjects who received at least one dose of IMC-CS4 will be included in the Safety Population, regardless of their eligibility for the study. The Safety population will be used for the analysis of baseline characteristics, efficacy data and safety data.

# 5.1.3 Maximum Tolerated Dose Limiting Toxicity (MTDDLT) Population

Subjects who complete the initial 6 weeks of therapy<sup>1</sup> or experience a DLT during the first cycle will be included in the MTD-DLT Population. Patients who discontinued during the initial 6 weeks due to reasons other than DLT will be excluded from the MTD DLT population. The MTD-DLTD population will be used for the evaluation of DLTs in order to determine the MTDRP2D.

#### 5.2 Definitions and data handling conventions

#### 5.2.1 Safety Data Handling and Definitions

### **5.2.1.1 Coding**

Adverse events: All adverse events (AE) will be coded by the Medical
Dictionary for Regulatory Activities (MedDRA<sup>TM</sup>) and graded according to the
National Cancer Institute (NCI) Common Terminology Criteria for Adverse
Events (CTCAE), Version 4.0 (version 4.0 includes all of the minor versions
4.0x).

<sup>&</sup>lt;sup>1</sup> i.e. first four infusions completed, plus an observation period of 21 days after last dose in cycle 1 or entry into cycle 2 if start of cycle 2 occurs before completion of the 21 days observation. IMC-CS4 (LY3022855)

 Pre treatment Therapy and Concurrent Therapy: Current medications, medications taken within 30 days prior to first dose of study therapy, prior cancer therapy will be coded using the WHOdrug.

## **5.2.1.2** Treatment-Emergent Adverse Events

An AE will be regarded as **treatment-emergent** if its onset date occurs any time after the administration of the first dose of study medication, up to 30 days after the last dose of study medication (or up to any time if related to study medication), or if it occurs prior to first dose date and worsens while on study medication.

#### 5.2.1.3 Partial Dates for Adverse Events, Concomitant Medications and Birthday

For the patient data listings no imputation of incomplete dates will be applied. The listings will show the incomplete dates without any change. Dates with missing day or both day and month, will adhere to the following conventions:

- The missing day of onset of an adverse event or start date of a concurrent therapy will be set to:
  - The date of the first study treatment, if the onset year and month is the same as year and month of the first study treatment
  - First day of the month that the event occurred, if the onset year and month is after the year and month of first study treatment
  - The date of informed consent, if the onset month/year is before the month/year of the first study treatment.
  - •\_\_\_
- If the onset date of an adverse event or start date of a concurrent therapy is missing both, day and month, the onset date will be set to:
  - The date of the first study treatment, if the onset year is the same as the year of the first study treatment
  - January 1 of the year of onset, if the onset year is after the year of the first study treatment

- The missing day of resolution of an adverse event or end date of a concurrent therapy will be set to the last day of the month of the occurrence. If the patient died the same month, then set the imputed date as the date of death.
- If the resolution date of an adverse event or end date of a concurrent therapy is missing both the day and month, the date will be set to:
  - December 31 of the year of occurrence. If the patient died the same year, then set the imputed date as the date of death.

Only year of birth is collected in the study. Age will be derived from year of birth by setting the date to 1 July of the year of birth.

#### 5.2.1.4 Study Drug Exposure

Exposure analyses will be based on the actual dose administered (in mg) and body weight (in kg) per the eCRF. The baseline body weight will be used for calculating the cumulative dose unless the subject's weight changes  $\geq 10\%$ . For subjects with a weight change  $\geq 10\%$ , the revised weight will be used from the time point of the change and onwards.

For analysis of dose exposure **across all cycles** the following definitions will be used:

- Duration of cycle:
  - Patients discontinuing during first cycle: Duration of cycles (in weeks)<sup>2</sup> = (Date of last dose date of first dose+21) / 7
  - Patients discontinuing treatment after start of Cycle 2: Duration of cycles (in weeks)<sup>3</sup> = (Date of last dose date of first dose+7) / 7
- Duration of treatment:
  - Patients discontinuing during first cycle: Duration of treatment (in weeks)<sup>4</sup> = (Date of last dose date of first dose+7) / 7

<sup>&</sup>lt;sup>2</sup> 21 days added to duration of cycle because of a 2 week observation period after last dose in cycle 1 (ie, 21 days until the next dose).

<sup>&</sup>lt;sup>3</sup> 7 days added to duration of cycle because administrations are planned every week (starting from Cycle 2).

<sup>&</sup>lt;sup>4</sup> 7 days added to duration of treatment because administrations are planned every week. Duration of treatment does not include the 2-week observation period in Cycle 1. IMC-CS4 (LY3022855)

- Patients discontinuing treatment after start of Cycle 2: Duration of treatment (in weeks)<sup>5</sup> = Duration of cycle -14
- Cumulative dose (mg/kg) = Sum of all [administered dosages (mg) / baseline weight<sup>6</sup> (kg)]
- Dose intensity (mg/kg/week) = Cumulative dose / Duration of treatment
- Planned weekly dose: Refer to Table 1: Planned Dose Regimens
- Relative dose intensity (%) = (Dose intensity / Planned weekly dose) \* 100.
- Number of dose reductions: total number of reduction steps comparing the intended dose level before each infusion (as entered in the eCRF) to the protocol planned dose level as referenced in Table 2: General Dose Reduction Guidelines.
- Dose delay within a cycle: a dose is considered delayed if it is administered more than 3 days after the scheduled date relative to the previous administration.

| Table 1: | Planned | Dose 1 | Regimens |
|----------|---------|--------|----------|
|----------|---------|--------|----------|

| Cohort | All cycles | Dosing Frequency |
|--------|------------|------------------|
| 1 | 2.5 mg/kg | Weekly |
| 2 | 0.3 mg/kg | Weekly |
| 3 | 0.6 mg/kg | Weekly |
| 4 | 1.25 mg/kg | Every 2 weeks |
| 5 | 1.25 mg/kg | Weekly |
| 6 | 2.5 mg/kg | Every 2 weeks |

For analysis of dose exposure **in Cycle 1 only** the same definitions as across all cycles will be used except the following:

Duration of cycles (in weeks)<sup>7</sup> = (Date of last dose – date of first dose+21) / 7
 Or if start of cycles 2<sup>8</sup> occurs before last dose of cycle 1 + 21 days:
 Duration of cycles (in weeks)= (Date of start Cycle 2-date of first dose)/7

IMC-CS4 (LY3022855)

<sup>&</sup>lt;sup>5</sup> 14 days is subtracted from the duration of cycle because the 2-week observation period is excluded from the duration of treatment.

<sup>&</sup>lt;sup>6</sup> Except in case of weight change from baseline ≥10% as described above.

<sup>&</sup>lt;sup>7</sup>21 days added to duration of cycle, because of a 2-week observation period after last dose in Cycle 1 (i.e. 21 days until the next dose).

<sup>&</sup>lt;sup>8</sup> Start of Cycle 2 is defined as day of first infusion of Cycle 2.

• Cumulative dose (mg/kg) = Sum of [all administered dosages during cycle 1 (mg) / baseline weight (kg)]

**Table 2: General Dose Reduction Guidelines** 

| Cohort | Planned Starting dose | First Reduction | Second Reduction |
|---|---|---|---|
| 1 | 2.5 mg/kg weekly | Discontinue IMC-CS4 | - |
| 2 | 0.3 mg/kg weekly | Discontinue IMC-CS4 | - |
| 3 | 0.6 mg/kg weekly | 0.3 mg/kg weekly | Discontinue IMC-CS4 |
| 4 | 1.25 mg/kg every 2 weeks | 0.6 mg/kg every 2 weeks | 0.3 mg/kg every 2<br>weeks |
| 5 | 1.25 mg/kg weekly | 0.6 mg/kg weekly | 0.3 mg/kg weekly |
| <u>6</u> | 2.5 mg/kg every 2 weels | 1.25 mg/kg every 2<br>weeks | 0.6 mg/kg every 2<br>weeks |

Note: Actual dose levels entered in the CRF will be rounded to the nearest dose level listed in this table (e.g. any IMC-CS4 dose level >5 and < 7.5 mg/kg will be rounded to 5 mg/kg for the purpose of the dose reduction calculation). No dose reductions are allowed after a DLT. In the setting of non-life-threatening reversible Grade ≤ 3 IMC-CS4-related toxicities that do not meet the definition of a DLT, IMC-CS4 may be held (if appropriate in the opinion of the Investigator) for a maximum of 3 weeks, until resolution to Grade < 2.

## **5.2.2 Efficacy Data Handling and Definitions**

Study evaluations will take place in accordance with the flow chart in Section 7.6 of the CP24-1001 Study Protocol.

Subjects will be evaluated for response according to RECIST 1.1 guidelines.[i] Subjects will be evaluated for response every 6 weeks (± 3 days) following the first dose of study therapy until radiographic documentation of PD, even if therapy is delayed due to toxicity or for other reasons.

#### **5.2.2.1 Determination of Best Overall Response (BOR)**

The Best Overall Response (BOR) will be determined using the RECIST (Version 1.1) guidelines. It is defined as the best response across all time points from the start of the treatment until disease progression based on investigators assessment. When SD is believed to be best overall response, it needs to be assessed a minimum of 39 days (ie, 6 weeks – 3 days as allowed per protocol) after start of treatment. Otherwise, the best overall response will be NE, unless any PD was further documented, in which case BOR will be PD. Tumor response (ie, for complete response [CR] or partial response [PR]) will not be confirmed following initial documentation of objective response.

## 5.2.3 General Data Handling

- Continuous variables will be summarized using descriptive statistics, ie, number
  of non-missing records (n), mean, median, standard deviation, minimum, and
  maximum.
- Categorical variables will be summarized by frequency and its corresponding percentage.
- Missing Data: All analyses and descriptive summaries will be based on the observed data. Unless otherwise specified, missing data will not be imputed or "carried forward."
- **Baseline Measurement**: Unless otherwise specified, the last valid (ie, non-missing) measurement prior to the first dose of study medication will serve as the baseline measurement.
- **Date of Birth**: CRF records only the year of birth. For analysis purposes, July 1 will be used as the month and day of birth
- Age (years) = (Date of informed consent Date of birth + 1) / 365.25
- **Duration**: Duration is calculated as:
  - Duration (days) = (End Date Start Date + 1)
  - Duration (weeks) = (End Date Start Date + 1) / 7

- Duration (months) =  $(\text{End Date} \text{Start Date} + 1) / 30.4375^9$
- Duration (years) =  $(\text{End Date} \text{Start Date} + 1) / 365.25^{10}$

#### 5.3 Data analysis

## **5.3.1** Disposition of Patients

The number of patients enrolled and the number of screening failures will be presented. Number (percent) of patients who were in the Safety population and in the MTD-DLT population, discontinued treatment and discontinued study as of data cut-off date will be summarized. A patient will be considered as off treatment if the End of Treatment form has been completed. A patient will be considered as off study if the End of Study visit has been completed or withdrew consent (ie, discontinued treatment due "withdrawal of consent" according to the End of Treatment form). Number (percent) of patients who discontinued will also be summarized by reason for discontinuation. A listing of patients with protocol deviations will be provided.

# **5.3.2 Demographic and Baseline Characteristics**

The following demographic and baseline characteristics will be summarized using the Safety population:

## Demographic:

- Age (years) and age categories (<65 years vs. ≥65 years)
- Gender
- Race and Ethnicity
- Height (cm)
- Weight (kg)
- Eastern Cooperative Oncology Group (ECOG) performance status

<sup>&</sup>lt;sup>4</sup>Days in months = average number of days in a year / 12.

<sup>&</sup>lt;sup>5</sup>Average number of days in a year = 365.25, reflecting the Julian Year of three years with 365 days each and one leap year of 366 days.

IMC-CS4 (LY3022855)

#### Medical history

Pre-treatment disease characteristics:

- Cancer type
- Initial and current TNM staging
- Pathological confirmation of malignancy
- Sites of Metastatic Disease
- Duration of disease (months from pathological confirmation of malignancy to first dose; if the day of confirmation of malignancy is unknown it will be replaced by 15MMMYYYY)

Prior anticancer treatments or surgery:

- Type of therapy
- Prior Surgery

Baseline vital signs, physical examination, laboratory assessments, tumor assessments will be included in the tables summarizing these variables across scheduled study visits.

#### 5.3.3 Analysis of Efficacy Data

Efficacy data will be analyzed overall using the Safety population.

#### **5.3.3.1** Response

Best overall response rate (number of subjects who achieve a best response of CR or PR during therapy divided by the total number of subjects treated) and disease control rate (number of subjects who achieve a best response of CR or PR or SD during therapy divided by the total number of subjects treated) will be presented for each cohort of subjects and overall. In addition all tumor assessments will be included in patient listings.

#### 5.3.4 Analyses of Safety Data

#### 5.3.4.1 Study Drug Exposure

The following variables will summarized according to the definitions provided in section 5.2.1.4. Exposure analyses will include the following:

## Cycle 1 only using the MTD population:

- Number of infusions
- Cumulative dose (mg/kg)
- Dose intensity (mg/kg/week)
- Adjusted dose intensity (mg/kg/week)
- Relative dose intensity (%)
- Number (%) of subjects with dose modifications (reduced or change of infusion rate).

#### Across all cycles using the Safety population

- Duration of treatment (weeks)
- Duration of cycles (weeks)
- Number (%) of subjects treated by cycle.
- Number of infusions
- Cumulative dose (mg/kg)
- Dose intensity (mg/kg/week)
- Adjusted dose intensity (mg/kg/week)
- Relative dose intensity (%)
- Number (%) of subjects with dose modifications (reduced or change of infusion rate).

#### 5.3.4.2 Dose Delays and Dose Modifications

The number and percentage of patients with dose delays > 3 days (within Cycle 1 and overall) will be presented. The number and percentage of patients with any dose reduction (reduction to first or second dose level) will also be presented. IMC-CS4 (LY3022855)

Version 2.0

#### 5.3.4.3 Treatment Emergent Adverse events

Treatment-emergent AEs will be summarized by MedDRA® System Organ Class (SOC) and preferred term (PT), classified from verbatim terms. The incidence and percentage of subjects with at least one occurrence of a preferred term will be included, according to the most severe NCI-CTCAE grade. Causality (relationship to study drug) will be summarized separately. If more than one AE is recorded for a patient within any SOC or PT term, the patient will only be counted once on the most severe grade and the closest relationship to treatment.

AEs reported with a causal relationship of 'possiblye related' and 'probablye related' to study medication or 'does not know' will be considered related to study medication.

Missing classifications concerning study medication relationship will be considered as related to study medication.

The following will be summarized using the Safety population for all AEs, and the MTD population for AEs with onset date in Cycle 1 (ie, within 21 days after last dose in Cycle 1 and prior to start of Cycle 2):

- All AEs,
- SAEs,
- NCI-CTCAE Grade 3 or higher AEs,
- Related AEs, SAEs, and NCI-CTCAE Grade 3 or higher AEs,
- AEs leading to dose modification, study medication discontinuation, and death will be summarized according to MedDRA® Preferred Terms.
- Duration of AE will be determined and included in listings along with action taken and outcome.

#### **5.3.4.4 Dose-Limiting toxicity**

The number of subjects who experience any DLT during Cycle 1 (ie, within 21 days after last dose in Cycle 1 and prior to start of Cycle 2) will be presented based on all DLT-evaluable subjects (MTD population).

#### 5.3.4.5 Death

All deaths that occur within 30 days of last dose of study medication as well as cause of death will be listed using the Safety population.

# 5.3.4.6 Performance Status, Physical Exams, Vital Signs, ECG and Laboratory Evaluations

#### 5.3.4.6.1 Laboratory Evaluation

Laboratory results will be classified according to NCI-CTCAE grade. Laboratory results not corresponding to an NCI-CTCAE term will not be graded. Laboratory toxicity shifts from baseline to worst grade will be provided. The last measurement before study medication will serve as the baseline measurement. Results for variables that are not part of the NCI-CTCAE will be presented in the listings as below, within, or above the normal limits of the local laboratory.

#### 5.3.4.6.2 ECOG Performance status, Physical Exams and ECG

The results from physical examination, ECOG performance status and ECG will be tabulated.

The frequency of physical examination abnormalities will be summarized by scheduled time point.

ECOG performance status will be presented in a shift table.

Additionally, the frequency of abnormal ECG parameters will be tabulated by scheduled time point.

#### **5.3.4.6.3** Vital signs

Vital sign measurements will be summarized using the following categories:

IMC-CS4 (LY3022855)

Version 2.0

- Body Temperature (C):  $<36, 36-38.5, \ge 38.5$
- Systolic Blood Pressure (mmHg): <140, 140-160, ≥160
- Diastolic Blood Pressure (mmHg): <90, 90-100, ≥100
- Arterial Pulse (beats/min):  $<60, 60-120, \ge 120$
- Respiratory Rate (breaths/min):  $\langle 20, 20\text{-}30, \geq 30 \rangle$

Vital signs will be obtained weekly during the Treatment period. At every visit that includes administration of study medication, vital signs to be checked and recorded prior to each infusion of IMC-CS4, midway through each infusion, at the end of each infusion, and every 15 minutes for the first hour following each infusion

Pre-infusion and post-infusion measurements at each visit will be presented as shift tables from:

- Preinfusion to Highest-on-Infusion
- Preinfusion to Lowest-on-Infusion
- Preinfusion to End-of-Infusion

#### **5.3.5** Other Assessments or Analyses

#### 5.3.5.1 Pharmacokinetic Assessments

Blood samples for PK will be analyzed by the ImClone Department of Clinical Pharmacology. Parameters to be reported may include, but not be limited to,  $C_{max}$ ,  $C_{min}$ , AUC,  $t_{1/2}$ , Cl, and  $V_{ss}$  of IMC-CS4, and will be generated using a noncompartmental model. PK parameters will be summarized using descriptive statistics.

#### **5.3.5.2** Pharmacodynamic Assessments

Tissue (DNA, RNA and protein analyses) and whole blood analyses, including analyses of circulating levels of CSF-1, will be descriptive, and correlations to safety and/or

IMC-CS4 (LY3022855)

efficacy will be performed as appropriate. <u>There will be a separate SAP describing the analysis of pharmacodynamic assessments.</u>

# 5.4 Interim analyses and data monitoring committees

For more details about safety reviews and monitoring committees please refer to Section 12.6.28 of the protocol.

# 5.5 Changes in planned analyses from the protocol

None

# 6 Planned summary tables and Listings

Planned table numbering and title may be modified for the clinical study report (CSR), with the final list to be reflected in a separate table shell document.

# **6.1 Planned Demographic Tables**

| Table | Table Title | Population |
|--------|------------------------------------------|--------------|
| Number | | |
| 14.1.1 | Patient Disposition | All enrolled |
| | | patients |
| 14.1.2 | Demographic and Baseline Characteristics | Safety |
| 14.1.3 | Pre-Treatment Disease Characteristics | Safety |
| 14.1.4 | Sites of Metastatic Disease at Screening | Safety |
| 14.1.5 | Prior Anti-Cancer Therapy or Surgery | Safety |
| 14.1.6 | Medical History | Safety |

# **6.2 Planned Efficacy Tables**

| Table | Table Title | Population |
|---|---|---|
| Number | | |
| 14.2.1 | Best Overall Response, Disease Control Rate and Response | Safety |
| | Rate | |

# **6.3 Planned Safety Tables**

| Table | Table Title | Population |
|---|---|---|
| Number | | |
| | Dose Exposure | |
| 14.3.1.1 | IMC-CS4 Dose Exposure in Cycle 1 | DLT |
| 14.3.1.2 | IMC-CS4 Dose Exposure | Safety |
| 14.3.2 | IMC-CS4 Dose Delays and Modifications in Cycle 1 | DLT |
| 14.3.2 | IMC-CS4 Dose Delays and Modifications | Safety |
| | Adverse events | |
| 14.3.5 | Summary of Adverse Events | Safety |
| 14.3.6 | DLTs by SOC and PT (Cycle 1) | DLT |
| 14.3.7.1 | Adverse Events by SOC and PT | Safety |
| 14.3.7.2 | Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.8.1 | Severe Adverse Events by SOC and PT | Safety |
| 14.3.8.2 | Severe Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.9.1 | Serious Adverse Events by SOC and PT | Safety |
| 14.3.9.2 | Serious Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.10.1 | Related Adverse Events by SOC and PT | Safety |
| 14.3.10.2 | Related Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.11.1 | Related Severe Adverse Events by SOC and PT | Safety |
| 14.3.11.2 | Related Severe Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.12.1 | Related Serious Adverse Events by SOC and PT | Safety |
| 14.3.12.2 | Related Serious Adverse Events by SOC and PT (Cycle 1) | DLT |
| 14.3.13.1 | Adverse Events Resulting in Treatment Delay or Modifications by SOC and PT | Safety |
| 14.3.13.2 | Adverse Events Resulting in Treatment Delay or Modifications by SOC and PT (Cycle 1) | DLT |

IMC-CS4 (LY3022855)

Version 2.0

| 14.3.14.1 | Adverse Events Resulting in Treatment Discontinuation by SOC and PT | Safety |
|---|---|---|
| 14.3.14.2 | Adverse Events Resulting in Treatment Discontinuation by SOC and PT (Cycle 1) | DLT |
| 14.3.15.1 | Adverse Events Resulting in Death by SOC and PT | Safety |
| 14.3.15.2 | Adverse Events Resulting in Death by SOC and PT (Cycle 1) | DLT |
| 14.3.16.1 | Adverse Events by SOC and PT and Worst Grade | Safety |
| 14.3.16.2 | Adverse Events by SOC and PT and Worst Grade (Cycle 1) | DLT |
| 14.3.17 | Deaths | Safety |
| | Physical Examination, Vital Signs, Laboratory Assessments, ECG | |
| 14.3.18 | Physical Examination Abnormalities by Scheduled Time | Safety |
| 14.3.19 | ECOG Performance Status Shift Table | Safety |
| 14.3.20.3 | Vital Signs Shift from Pretreatment to End-of-Study | Safety |
| 14.3.21.1 | Vital Signs Shift from Preinfusion to Highest-on-Infusion | Safety |
| 14.3.21.2 | Vital Signs Shift from Preinfusion to Lowest-on-Infusion | Safety |
| 14.3.21.3 | Vital Signs Shift from Preinfusion to End-of-Infusion | Safety |
| 14.3.22.1 | Laboratory CTC Grade Shift from Baseline to Worst Post Baseline Grade- Tests Graded in Single Direction(Either Above or Below Normal Range) | Safety |
| 14.3.22.2 | Laboratory CTC Grade Shift from Baseline to Worst Post Baseline<br>Grade- Tests Graded in Single Direction(Either Above or Below<br>Normal Range) | Safety |
| 14.3.22.3 | Laboratory CTC Grade Shift from Baseline to Worst Low Post Baseline<br>Grade -Tests Graded in Both Directions (Above and Below Normal<br>Range) | Safety |
| 14.3.23 | Laboratory CTC Grade Shift Shift from Pretreatment to End-of-Study | Safety |
| 14.3.24 | Electrocardiogram | Safety |
| 14.3.25 | Pharmacodynamic Biomarkers | Safety |
| 14.3.26 | IMC-CS4 Antibodies | Safety |

# **6.4 Planned Patient Data Listings**

| Listing | Listing Title | Population |
|---------|------------------------------------------|-----------------------|
| Number | | |
| | Baseline Characteristics | |
| 1 | Patient Disposition | All enrolled patients |
| 2.1 | Definition of In- and Exclusion Criteria | NA |
| 2.2 | Inclusion Criteria | All enrolled patients |
| 2.3 | Exclusion Criteria | All enrolled patients |
| 2.4 | Exemption of In- and Exclusion Criteria | All enrolled patients |
| 3 | Protocol Deviations | Safety |
| 4 | Demographic and Baseline Characteristics | Safety |
| 5 | Pre-Treatment Disease Characteristics | Safety |
| 6 | TNM Staging | Safety |
| 7 | Site of Metastatic Disease at Screening | Safety |
| 8 | Previous Anti-Cancer Therapy | Safety |
| 9 | Prior Disease Related Radiotherapy | Safety |
| 10 | Prior Disease-Related Surgery | Safety |
| 11 | Medical History | Safety |
| 12 | Pregnancy Test | Safety |
| | Efficacy | |
| 13.1 | Tumor Measurements – Target Lesions | Safety |
| 13.2 | Tumor Measurements – Non-Target Lesions | Safety |
| 13.3 | Tumor Measurements – New Lesions | Safety |
| 13.4 | Tumor Measurements – Comments | Safety |
| 13.5 | Best Overall Response | Safety |
| 13.6 | Radiographic Scans | Safety |
| | Dose Exposure | |
| 14.1 | IMC-CS4 Administration | Safety |
| 14.2 | IMC-CS4 Modifications | Safety |
| 14.3 | IMC-CS4 Infusion Interruptions | Safety |

IMC-CS4 (LY3022855)

Version 2.0

| 14.4 | IMC-CS4 Dose intensity | Safety |
|---|---|---|
| | Adverse Events | |
| 15.1 | Dose-Limiting Toxicities | DLT |
| 15.2 | Adverse Events | Safety |
| 15.3 | Serious Adverse Events | Safety |
| 15.4 | Adverse Events Resulting in IMC-CS4 Modifications | Safety |
| 15.5 | Adverse Events Resulting in IMC-CS4 Treatment Discontinuation | Safety |
| 15.6 | Adverse Events Resulting in Death | Safety |
| 15.7 | Adverse Event Comments | Safety |
| 16.1 | Concurrent Therapy and Procedures for the Treatment of AEs | Safety |
| 16.2 | Concurrent Therapies and Procedures not for the Treatment of AEs | Safety |
| 17 | Death Reports | Safety |
| | Physical Examination, Vital Signs, Laboratory Assessments | |
| 18 | Weight, Height and ECOG Performance Status | Safety |
| 19 | Physical Examination | Safety |
| 20 | Vital Signs | Safety |
| 21.1 | Laboratory Reference Ranges | NA |
| 21.2 | Listing of Patients With ≥Grade 3 Abnormal Laboratory Results | Safety |
| 22 | Laboratory - Hematology | Safety |
| 23 | Laboratory - Coagulation | Safety |
| 24 | Laboratory - Serum Chemistry | Safety |
| 25 | Laboratory - Urinanalysis | Safety |
| 26 | Electrocardiogram | Safety |
| 27 | Hospitalization | Safety |
| 28 | Pharmacodynamic Biomarkers | Safety |
| 29 | IMC-CS4 Antibodies | Safety |

## **Appendix 1: List of Abbreviations**

AE adverse event

BOR best overall response CR complete response

CRO contract research organization CSF-1 colony-stimulating factor-1

CSF-1R colony-stimulating factor-1 receptor

CSR Clinical study report
DLT dose-limiting toxicity
ECG electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF electronic case report form

FPV first patient visit

MedDRA<sup>®</sup> Medical Dictionary for Regulatory Activities

MTD maximum tolerated dose

NCI-CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NE non-evaluable
PD progressive disease
PK pharmacokinetic(s)
PR partial response
PT preferred term

RECIST 1.1 Response Evaluation Criteria in Solid Tumors, Version 1.1

SAE serious adverse event SAP Statistical Analysis Plan

SD stable disease SOC system organ class

TNM tumor, nodes, and metastases

WHOdrug world health organization drug information

# **Appendix 2: References**

i Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). European Journal of Cancer. 2009;45:228-247.

Leo Document ID = 312596ef-b316-45fd-85f3-21975686e318

Approver: PPD

Approval Date & Time: 19-Oct-2012 17:39:32 GMT Signature meaning: Approved